CLINICAL TRIAL: NCT03567798
Title: A Post Marketing Randomized Placebo Controlled Study to Evaluate the Efficacy of Study Product UPLAT® (Carica Papaya Leaf Extract + Tinospora Cardifolia Extract) in the Cancer Patients With Thrombocytopenia Induced by Chemotherapy
Brief Title: Thrombocytopenia Induced by Chemotherapy
Acronym: papayaleaf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Socrates School Of Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPL/UP/2017/01
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Intervention Model Description: Single blind, randomized, multicentric placebo controlled study
Who Masked: Participant
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): UPLAT® (Carica papaya leaf Extract + Tinospora cardifolia Extract
  Take 4 units daily (2 in morning and 2 in evening) for 10 days
  Interventions: Dietary Supplement: UPLAT
- B (Placebo Comparator): Placebo
  Take 4 units daily (2 in morning and 2 in evening) for 10 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: UPLAT — Carica papaya leaf Extract + Tinospora cardifolia Extract
  Arms: A
Other: Placebo — Placebo
  Arms: B

SUMMARY:
Single blind, randomized, multicentric placebo controlled study to evaluate the efficacy of Study product in patient with Chemotherapy induced thrombocytopenia. The Study is divided into [screening visit (visit 1) > baseline and treatment allocation visit (visit 2) >blood collection (visit 3); treatment compliance visit (visit 4) > blood collection (visit 5) >blood collection (visit 6)>end of study visit (visit 7)].

DETAILED DESCRIPTION:
UPLAT® (Carica papaya leaf Extract + Tinospora cardifolia Extract), is an orally administered dietary supplement for management of thrombocytopenia. Manufactured bySanat Products Ltd.

Throughout study, it will be designated as product A to maintain study blindness at subject end.

Placebo Throughout study, it will be designated as product B to maintain study blindness at subject end.

Single blind, randomized, multicentric placebo controlled study to evaluate the efficacy of Study product in patient with Chemotherapy induced thrombocytopenia. The Study is divided into [screening visit (visit 1) > baseline and treatment allocation visit (visit 2) >blood collection (visit 3); treatment compliance visit (visit 4) > blood collection (visit 5) >blood collection (visit 6)>end of study visit (visit 7)].

Dose regimen After meeting the inclusion criteria subject will take 4 units daily (2 in morning and 2 in evening) for 10 days. Patients will be called on Day5th, 10th and 15thfor the Complete blood count (Central lab).

Total blood loss Approximately 8-12 mL

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18-55 years.
2. Subjects must sign with date an informed consent prior to any evaluation and participation in the trial.
3. Patients who were confirmed solid tumour and received at least one cycle of chemotherapy prior to screening visit.
4. Patients with a platelet counts between > 20000 and < 150,000/ml at the time of screening.

Exclusion Criteria:

1. Planning to receive any type of surgery.
2. Pregnant or lactating women.
3. Patients with platelet count less than 20000/ml.
4. Patients with thrombocytopenia presenting with active bleeding.
5. Patients who have received blood or blood product transfusion during the current illness or during past one week.
6. Patients with thrombocytopenia purpura (ITP) leukemia, hemophilia or bleeding diathesis.
7. Participation in another trial with another investigational product

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Increase in the platelet counts from baseline levels to the end of therapy. | Day 15
  Increase in the platelet counts from baseline levels to the end
  of therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- North East Cancer Centre Hospital and research Institute, Guwahati, Assam, India

IPD SHARING:
Plan to Share IPD: Undecided
Not Yet Decided